CLINICAL TRIAL: NCT01957488
Title: Investigating the Safety and Performance of Two New 1-piece Ostomy Products in 180 Subjects With Ileostomy
Brief Title: Investigating the Safety and Performance of Two New 1-piece Ostomy Products Compared With SenSura 1-piece
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CP242
Record Dates: First submitted 2013-08-06; First posted 2013-10-08 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-08

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment sequence 1; First Coloplast Test product 1 (Experimental): The subjects are randomised 1:1:1 into six possible treatment groups to ensure random allocation of treatment to periods.
  Subjects are first allocated to test Coloplast Test product 1 and secondly test either:
  1. Coloplast Test product 1 and thereafter Coloplast SenSura
  2. Coloplast Sensura and thereafter Coloplast Test product 2
  Interventions: Device: Coloplast Test Product 1; Device: Coloplast Test Product 2; Device: Coloplast SenSura
- Treatment seqence 2; First Coloplast Test product 2. (Experimental): The subjects are randomised 1:1:1 into six possible treatment groups to ensure random allocation of treatment to periods.
  Subjects are first allocated to test Coloplast Test product 2 and secondly test either:
  1. Coloplast Test product 1 and thereafter Coloplast SenSura
  2. Coloplast Sensura and thereafter Coloplast Test product 1
  Interventions: Device: Coloplast Test Product 1; Device: Coloplast Test Product 2; Device: Coloplast SenSura
- Treatment sequence 3, First Coloplast SenSura (Experimental): The subjects are randomised 1:1:1 into six possible treatment groups to ensure random allocation of treatment to periods.
  Subjects are first allocated to test Coloplast SenSura and secondly test either:
  1. Coloplast Test product 2 and thereafter Coloplast Test product 1
  2. Coloplast Test product 1 and thereafter Coloplast Test product 2
  Interventions: Device: Coloplast Test Product 1; Device: Coloplast Test Product 2; Device: Coloplast SenSura

INTERVENTIONS:
Device: Coloplast Test Product 1 — Coloplast Test product 1 is a newly developed 1-piece ostomy appliance
Device: Coloplast Test Product 2 — Coloplast Test product 2 is a newly developed 1-piece ostomy appliance
Device: Coloplast SenSura — SenSura 1-piece is the commercial available CE-marked SenSura 1-piece from Coloplast A/S.
  Other Names: SenSura 1-piece

SUMMARY:
The aim of the current investigation is to investigate the performance of two new 1-piece ostomy products

DETAILED DESCRIPTION:
The present investigation aims at testing the performance and safety of the two new 1-piece ostomy products

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent and signed letter of authority (mandatory in DK)
2. Be at least 18 years of age and have full legal capacity.
3. Be able to handle the products themselves
4. Have an ileostomy with a diameter between 10 and 40 mm.
5. Have had their ostomy for at least three months.
6. Have within the last month used a 1-piece flat product with open bag
7. Currently using midi or maxi bags
8. Willing to use minimum 1 product every second day, i.e. maximum 2 days wear time.
9. Be suitable for participation in the investigation
10. Must be able to use custom cut product
11. Negative result of a pregnancy test for women of childbearing age (only DK)

Exclusion Criteria:

1. Currently receiving or have within the past 2 months received radio- and/or chemotherapy.
2. Currently receiving or have within the past month received systemic steroid or local treatment in the peristomal area
3. Are pregnant or breastfeeding
4. Participating in other interventional clinical investigations or have previously participated in this investigation
5. Has participated in the previous explorative Coloplast studies CP236 and CP237
6. Are currently or during the study using ostomy belt
7. Has a stoma below skin surface
8. Currently suffering from peristomal skin problems (i.e.bleeding and/or broken skin)
9. Has known hypersensitivity towards any of the test products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birte P Jakobsen, MD, Principal Investigator — Coloplast A/S
Locations (4):
- Holtedam 3, Humlebæk, Denmark
- QPS Nederlands, Groningen, Netherlands
- Sykepleierklinikken, Larvik, Norway
- Synexus Limited, Chorley, Lancashire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were recruited through the Coloplast database and hospital sites.
Groups:
- SenSura/Test 1/Test 2: The subjects in this group test the following in the order described below:
  1. SenSura (the comparator)
  2. Test 1
  3. Test 2
  The products are single use products which in average are removed and re-applyed every1-2nd day.
- SenSura/Test 2/Test 1: The subjects in this group test the following in the order described below:
  1. SenSura (the comparator)
  2. Test 2
  3. Test 1
  The products are single use products which in average are removed and re-applyed every1-2nd day.
- Test 1/SenSura/Test 2: The subjects in this group test the following in the order described below:
  1. Test 1
  2. SenSura (the comparator)
  3. Test 2
  The products are single use products which in average are removed and re-applyed every1-2nd day.
- Test 1/Test 2/SenSura: The subjects in this group test the following in the order described below:
  1. Test 1
  2. Test 2
  3. SenSura (the comparator)
  The products are single use products which in average are removed and re-applyed every1-2nd day.
- Test 2/SenSura/Test 1: The subjects in this group test the following in the order described below:
  1. Test 2
  2. SenSura (the comparator)
  3. Test 1
  The products are single use products which in average are removed and re-applyed every1-2nd day.
- Test 2/Test 1/SenSura: The subjects in this group test the following in the order described below:
  1. Test 2
  2. Test 1
  3. SenSura (the comparator)
  The products are single use products which in average are removed and re-applyed every1-2nd day.
Period: Test Period 1 (2 Weeks)
Arm/Group | SenSura/Test 1/Test 2 | SenSura/Test 2/Test 1 | Test 1/SenSura/Test 2 | Test 1/Test 2/SenSura | Test 2/SenSura/Test 1 | Test 2/Test 1/SenSura
Started | 30 | 31 | 30 | 32 | 30 | 30
Completed | 27 | 28 | 26 | 29 | 27 | 24
Not Completed | 3 | 3 | 4 | 3 | 3 | 6
Not completed — Lost to Follow-up | 2 | 0 | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 2 | 1 | 0 | 3
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 2
Not completed — subject did not want to wait for cut bag | 0 | 0 | 0 | 0 | 1 | 0
Not completed — screen failure | 0 | 0 | 0 | 0 | 0 | 1
Period: Test Period 2 (2 Weeks)
Arm/Group | SenSura/Test 1/Test 2 | SenSura/Test 2/Test 1 | Test 1/SenSura/Test 2 | Test 1/Test 2/SenSura | Test 2/SenSura/Test 1 | Test 2/Test 1/SenSura
Started | 27 | 28 | 26 | 29 | 27 | 24
Completed | 24 | 27 | 25 | 28 | 25 | 23
Not Completed | 3 | 1 | 1 | 1 | 2 | 1
Not completed — Protocol Violation | 2 | 0 | 1 | 1 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Discontinue due to personal problems | 0 | 0 | 0 | 0 | 0 | 1
Period: Test Period 3 (2 Weeks)
Arm/Group | SenSura/Test 1/Test 2 | SenSura/Test 2/Test 1 | Test 1/SenSura/Test 2 | Test 1/Test 2/SenSura | Test 2/SenSura/Test 1 | Test 2/Test 1/SenSura
Started | 24 | 27 | 25 | 28 | 25 | 23
Completed | 23 | 26 | 25 | 28 | 25 | 23
Not Completed | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Of the183 randomised subjects 4 subjects were not exposed to a product and were only included in the safety population (N =179). Of the 179 subjects 5 subjects were not included in the ITT population as no endpoint data was recorded for these subjects. The ITT population consisted of 174 subjects. Baseline data is only summerized for ITT subjects.
Arm/Group | All Subjects
Number analyzed (Participants) | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 103

OUTCOME MEASURES:

1. Primary Outcome: Leakage
Description: The fraction of baseplates with No leakage/seeping under the baseplate was measured. Leakage/seeping under the baseplate was assessed after each baseplate change.
Time Frame: 14 +- 1 days
Measure: Number; unit: percentage of baseplates
Units Other Than Participants: baseplates
Groups:
- Test 1: Fraction of baseplates with No leakage/seeping under the baseplate for subjects testing Coloplast Test 1
- Test 2: Fraction of baseplates with No leakage/seeping under the baseplate for subjects testing Coloplast Test 2
- SenSura: Fraction of baseplates with No leakage/Seeping under the baseplate for subjects testing SenSura
Arm/Group | Test 1 | Test 2 | SenSura
Number analyzed (Participants) | 160 | 160 | 159
Number analyzed (baseplates) | 1867 | 1907 | 1933
percentage of baseplates | 50 | 61 | 59

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during each test period 2 weeks +- 1 day
Groups:
- Test 1: Subjects testing Coloplast Test 1
- Test 2: Subjects testing Coloplast Test 2
- SenSura: Subjects testing SenSura
Arm/Group | Test 1 | Test 2 | SenSura
Serious Adverse Events (participants affected / at risk) | 3/162 | 2/163 | 5/163
Other Adverse Events (participants affected / at risk) | 38/162 | 24/163 | 27/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test 1 (N=162) | Test 2 (N=163) | SenSura (N=163)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — not related to device
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to device
Superficial Abscess - surcically drained (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Unlikely related to device
Dehydration after abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Not related to device
Nephrolitiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to device
AC Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device
Blocked Stoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device
Lung Cancer Complication (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to device
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Unlikely related to device
Lacerations left hand requiring suturs following dog attack (Social circumstances) | 0 (0) | 0 (0) | 1 (1) — Not related to device
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test 1 (N=162) | Test 2 (N=163) | SenSura (N=163)
Skin irritation (Skin and subcutaneous tissue disorders) | 38 (54) | 24 (39) | 27 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes